CLINICAL TRIAL: NCT05583240
Title: Influence of Olfaction Essential Oils on the Consumption of Benzodiazepine Receptor Agonists & Z-Drugs (BZRAs) Prescribed as " if Needed " in Psychiatric Outpatients (HECBA-PSY).
Acronym: HECBA-PSY
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Etablissement Public de Santé Barthélemy Durand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21P01; 2019-A02345-52 (Registry Identifier: ANSM)
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Psychiatric Disorder; Benzodiazepine Withdrawal
Keywords: Essential Oil; Psychiatry; Olfaction; Anxiety; Insomnia
MeSH Terms: conditions — Mental Disorders; Anosmia; Anxiety Disorders; Sleep Initiation and Maintenance Disorders | interventions — Oils, Volatile

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Essential Oils (Experimental)
  Interventions: Drug: Essences and Essential Oils

INTERVENTIONS:
Drug: Essences and Essential Oils — Participants will received Essential Oils through a nasal stick during 4 weeks.

SUMMARY:
The goal of this interventional study is to test the use of olfactory Essential Oils through a nasal stick as one of the non-medicinal strategies to propose to the patient to reduce the consumption of medication in a population of stabilized patients with psychiatric disorder.

The main objective is to evaluate whether the olfaction of a mixture of essential oils can reduce the intake of BZRAs, prescribed if needed.

The investigators want to compare the number of medications prescribed on "if needed" basis before and after the introduction of Essential Oils.

A period prior to inclusion is used to assess the participant's frequency of BZRA use. Then, participants will received Essential Oils through a nasal stick during 4 weeks. During this period, the patient completes weekly anxiety and sleep scales and at the final visit, weekly and monthly anxiety and sleep scales.

DETAILED DESCRIPTION:
It is a common in psychiatry for a physician to prescribe a patient, regardless of pathology, a treatment to be taken punctually in case of anxiety, nervousness, irritability or difficulty falling asleep. This "if needed" treatment can be add to the patient's usual treatment or constitute his only drug treatment.

Most of the time, the "if needed" medication prescribed is a BZRA, which exposes the patient to the risk of creating dependency and drug abuse if the doses are multiplied.

In this context, it seems interesting to us to test the use of olfactory Essential Oils through a nasal stick as one of the non-medicinal strategies to propose to the patient to reduce the consumption of medication.

A two-week period prior to inclusion is used to assess the patient's frequency of BZRA use.

During the pre-inclusion visit, the investigators explain the study protocol, the patient gives consent, and they are given a diary to record their BZRA use.

(one of the inclusion criteria is more than 3 and less than 21).

At the second visit, the patient fills out the anxiety and sleep questionnaire, the investigators perform an allergy test, and they receive an aromastick.

At following visits, the patient completes weekly anxiety and sleep scales and at the final visit, weekly and monthly anxiety and sleep scales.

ELIGIBILITY:
Inclusion Criteria:

* Adult without legal protection measures
* Ambulatory followed up
* Stabilised main psychiatric pathology
* Patient having had recourse between 3 and 21 times a week in the previous 14 days to a benzodiazepine or related treatment, for anxiolytic or hypnotic purposes, prescribed "if necessary" (on request)
* Patient who understand French both orally and in writing
* Patient who do not have an identified organic cause for their disorder
* Patient who be affiliated to a social security scheme
* Patient who have given their free and informed consent and signed the consent form

Exclusion Criteria:

* Patients with asthma or unstable epilepsy
* Pregnancy or breastfeeding
* EO allergies
* Patients having already a regular consumption of EO for the study indication
* Patients under guardianship or under reinforced guardianship

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-04-19 (Actual); Primary Completion 2023-04-18 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Number of medications prescribed | 4 weeks
  Compare the number of medications prescribed on "if needed" basis before and after the introduction of essential oils.

SECONDARY OUTCOMES:
Anxiety level | 4 weeks
  STAI (State Trait Anxiety Inventory) scale
Sleep level | 4 weeks
  Pittsburgh Sleep Quality Index (PSQI) scale

CONTACTS AND LOCATIONS:
Overall Officials: Christian Trichard, Principal Investigator — Etablissement Public de Santé Barthélemy Durand
Locations (1):
- Etablissement Public de Santé Barthélemy Durand, Étampes, France

IPD SHARING:
Plan to Share IPD: No